CLINICAL TRIAL: NCT07058558
Title: Increasing Knowledge, Reducing Risk: A Community- Integrated Nutrition Education Intervention to Prevent Type 2 Diabetes in Peel
Brief Title: Community-integrated Nutrition Education to Prevent Type 2 Diabetes in Peel
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Vasanti Malik, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 46464
Record Dates: First submitted 2025-06-06; First posted 2025-07-10 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: Peel; Portfolio Diet; Nutrition; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: One-group pretest-posttest design for implementation science involving:
  1. Participation in a 12-month nutrition education intervention to prevent type 2 diabetes.
  2. Assessing the effect of the intervention on changes in body weight (primary outcome), waist circumference, blood pressure and diet quality after 1 year from baseline using a one-group pretest-posttest design.
  3. Assessing the effect of the intervention on biomarkers of T2D risk (glucose, insulin, lipids, HbA1c) after 1 year compared to baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Twelve month lifestyle intervention comprised of nutrition education and community gardening based on the Portfolio Diet
  Interventions: Behavioral: Nutrition Education and Community Gardening

INTERVENTIONS:
Behavioral: Nutrition Education and Community Gardening — Participants will be presented with 16 nutrition education modules based on the Portfolio Diet, through group-based virtual sessions delivered by the investigators for one year. In addition, participants will take part in two community gardening sessions during growing season, and will grow Portfolio Diet foods such as eggplant, okra, and temperate climate fruit.

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of an intervention that delivers nutrition education based on the Portfolio Diet on type-2 diabetes (T2D) risk factors among adults who are without chronic conditions, who have overweight and a high waist circumference plus one self-reported T2D risk factor. The main questions it aims to answer include:

1. What are the barriers and facilitators for effective implementation of the nutrition education intervention?
2. What is the effectiveness of the intervention on T2D risk factors?
3. What are implementation strategies for scaling up the intervention?

Participants will participate in a 12-month lifestyle intervention comprised of nutrition education based on the Portfolio Diet that includes community gardening sessions. In addition, participants will take part in pre-implementation focus groups/interviews and post-implementation focus groups/interviews.

DETAILED DESCRIPTION:
Peel has one of the highest rates of type 2 diabetes (T2D) in Ontario. Individuals with T2D have a higher risk of cardiovascular diseases (CVD), kidney disease, lower limb amputation and vision loss compared to the general population. Excess body weight, poor diet, and physical inactivity are key contributors to T2D risk, and are influenced by many factors including structural inequities and our built and food environments. Specific contributors in Peel include an urban design that discourages walking and a high proportion of residents with ethnic backgrounds at higher risk for T2D. There is an urgent need for local and practical T2D prevention strategies in Peel to ensure the health and quality of life of its residents. A healthy diet and lifestyle are important factors for preventing chronic diseases such as T2D.

The Portfolio Diet (PD) is an evidence-based healthy eating plan that has shown clinically meaningful reductions in T2D and CVD risk factors such as cholesterol and blood pressure in randomized controlled trials. Several prospective cohort studies have also shown the positive impact of the PD on the incidence of T2D and CVD. Given the strong scientific evidence, the PD is recommended by Diabetes Canada, the Canadian Cardiovascular Society and Obesity Canada.

An app for the PD (PortfolioDiet.app) was recently developed by the investigators. However, a strategy to deliver the PD at the community level has yet to be designed and evaluated. An intervention (program) that delivers tailored nutrition education based on the PD has the potential to be a successful strategy to address the T2D burden in Peel. This intervention (program) could help reduce barriers to accessing and understanding nutrition and health information, which are key elements of T2D prevention. A critical step to ensuring the success of such an intervention (program) is engaging with community stakeholders to design an effective implementation strategy.

The overarching aim of the proposed project is to assess the effectiveness of an intervention (program) that delivers nutrition education based on the PD on T2D risk factors. To achieve this, the investigators have partnered with the Peel Food Action Council (PFAC) and will conduct formative work using Consolidated Framework for Implementation Research (CFIR) to inform the implementation strategy for the intervention (program). The investigators also plan to incorporate community gardening sessions into the intervention led by PFAC to reinforce the nutrition education and enhance participant engagement. Community gardening programs have emerged as a strategy to improve diet quality especially when paired with nutrition education. The research questions pertain to understanding the barriers and facilitators for successful implementation of the intervention (program), evaluating its effectiveness on T2D risk factors and identifying implementation strategies for scaling up.

The specific aims are:

Aim 1: To conduct pre-implementation focus groups and interviews with the target population to inform the design of the intervention and implementation strategy.

Aim 1.2: To evaluate the effectiveness of the design of the curriculum and nutrition education modules teaching the Portfolio Diet through questionnaires and small group discussions with adults at risk of T2D (i.e. target population).

Aim 2: To assess the effect of the intervention among individuals at risk for T2D on changes in body weight, waist circumference, blood pressure and diet quality after 1 year compared to baseline.

Aim 2.1: To assess the effect of the intervention on biomarkers of T2D risk (glucose, insulin, lipids, HbA1c) after 1 year compared to baseline.

Aim 3: To conduct post-implementation focus groups and interviews with participants to determine the effectiveness of the intervention implementation and gather insights for scaling up.

ELIGIBILITY:
Inclusion Criteria:

* Must be in their 40s or older
* Must be a resident in the Peel region of the Greater Toronto Area
* Must not have any chronic conditions (that will impact participation in study)
* Must be overweight, have a high waist circumference plus one self-reported T2D risk factor (e.g. family history, non-white ethnicity, high blood pressure, high blood cholesterol, prediabetes)
* Must have a risk score of 21 or above using the CANrisk T2D screening tool (https://health.canada.ca/apps/canrisk-standalone/pdf/canrisk-en.pdf)
* Must not be participating in another trial
* Must have access to a smartphone or internet. (For participants who wish to join the study but do not have home internet/smart phone, the investigators will provide resources to participants such as locations/hours of public libraries and community centres, where they could access internet and/or an electronic device (i.e computers) to participate in the study).

Exclusion Criteria:

* Under the age of 40
* Not a resident in the Peel region of the Greater Toronto Area
* Has chronic conditions (that will impact participation in study)
* Not overweight, does not have a high waist circumference plus one self-reported T2D risk factor (e.g. family history, non-white ethnicity, high blood pressure, high blood cholesterol, prediabetes)
* Does not have a risk score of 21 or above using the CANrisk T2D screening tool (https://health.canada.ca/apps/canrisk-standalone/pdf/canrisk-en.pdf)
* Participating in another trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Weight in kilograms | From baseline to 1 year after
  Changes in body weight. Weight and height will be combined to report BMI in kg/m^2.

SECONDARY OUTCOMES:
Waist circumference in centimeters | From baseline to 1 year after
  Waist circumference will be measured in centimetres using measuring tape.
Height in Centimetres | From baseline to 1 year after
  Height will be measured using a stadiometer. Height and weight will be combined to report BMI in kg/m^2
Diet quality | From baseline to 1 year after
  Changes in diet quality will be assessed according to adherence to the Portfolio Diet, measured using the Harvard Food Frequency Questionnaire and 3-Day Diet Records using the Keenoa App. The Portfolio Diet score will be used to measure adherence with a score range between 6 and 30. A higher score indicates higher consumption of foods recommended in the diet.
Insulin in pmol/L | From baseline to 1 year after
  Insulin will be measured through a lab test at LifeLabs. A blood sample will be drawn by a healthcare professional and analyzed.
Glycated hemoglobin (HbA1c) as a percentage | From baseline to 1 year after
  Glycated hemoglobin (HbA1c) is a blood test that provides an average of blood sugar levels over the past 2-3 months. HbA1c will be measured through a lab test at LifeLabs. A blood sample will be drawn by a healthcare professional and analyzed.
Blood pressure (systolic pressure and diastolic pressure) | From baseline to 1 year after
  Both systolic pressure and diastolic pressure will be assessed for changes 1 year after baseline. Blood pressure will be measured using an automatic blood pressure machine.
Glucose Random in mmol/L | From baseline to 1 year after
  Glucose Random will be measured through a lab test at LifeLabs. A blood sample will be drawn by a healthcare professional and analyzed.
Lipids (Cholesterol/HDL/LDL/Triglycerides) in mmol/L | From baseline to 1 year after
  Lipid Profile, is a blood test that measures different types of lipids in blood, including cholesterol (total, HDL, and LDL) and triglycerides. This test will be done at Life Labs where a blood sample will be drawn by a healthcare professional and analyzed.
High-sensitivity C-reactive protein (hs-CRP) in mg/L | From baseline to 1 year after
  Hs-CRP is a marker of inflammation, and elevated levels can indicate increased cardiometabolic risk. A blood sample will be drawn by a healthcare professional at Life Labs and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Vasanti Malik, MSc, ScD, Principal Investigator — University of Toronto, Department of Nutritional Sciences; John Sievenpiper, MD, PhD, FRC, Study Chair — University of Toronto, Department of Nutritional Sciences; Laura Chiavaroli, MSc, PhD, Study Chair — University of Toronto, Department of Nutritional Sciences
Locations (2):
- Canada (2):
  - Community garden spaces across peel, Toronto, Ontario
  - University of Toronto Mississauga, Mississauga, Ontario (ON)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-05-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT07058558/ICF_000.pdf